CLINICAL TRIAL: NCT01673932
Title: Phase 1 Clinical Trial to Establish the Safety and Feasibility of Transplants of Umbilical Cord Blood Mononuclear Cells in Chronic Ischemic Stroke
Brief Title: Safety and Feasibility Study of Umbilical Cord Blood Mononuclear Cells Transplant to Treat Ischemic Stroke
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Spinal Cord Injury Network (Network)
Collaborators: Chinese University of Hong Kong (Other); The University of Hong Kong (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other); Queen Mary Hospital, Hong Kong (Other); StemCyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCB-IS-01
Record Dates: First submitted 2012-08-24; First posted 2012-08-28 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Stroke; Ischemic Stroke; Brain Ischemia
Keywords: stroke; chronic stroke; ischemic stroke; umbilical cord blood; mononuclear cell; transplant
MeSH Terms: conditions — Stroke; Ischemic Stroke; Brain Ischemia | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A - UCBMC Early Treatment Group (Experimental): Group A subjects will receive transplant of UCBMC isolated from HLA-matched umbilical cord blood at Day 0.
  Interventions: Biological: UCBMC; Procedure: surgery
- Group B - UCBMC Delayed Treatment Group (Experimental): Group B subject will partipate in 6 months observation and then receive the UCBMC transplant at month 6.
  Interventions: Biological: UCBMC; Procedure: surgery

INTERVENTIONS:
Biological: UCBMC — Transplant 10-40 million viable UCBMC suspension into brain adjacent to the infracted site
Procedure: surgery

SUMMARY:
The study is to assess the safety and possible efficacy of umbilical cord blood mononuclear cells (UCBMC) treatment of chronic ischemic stroke.

DETAILED DESCRIPTION:
This is an open-label, delayed-treatment trial.

A total of 12 subjects fulfill the inclusion and exclusion criteria will be recruited and randomly assigned into two treatment group. Group A (early-treatment group) will receive transplant of UCBMC isolated from HLA-matched umbilical cord blood at Day 0. Group B (delayed-treatment group) will participate in 6 months observation before the UCBMC transplantation at Month 6. All subjects will be followed up for 18 months from enrollment at Day 0. Long-term follow-up will be carried up to 36 months if applicable.

The adverse events and safety parameters will be collected and recorded. In addition, the stroke scores , gait and brain MRI will be obtained before and after the treatment to assess the safety and potential treatment effect of UCBMC in chronic ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* either gender, age 35 -65 years old;
* ischemic stroke > 6 months and < 60 months;
* stable hemiplegia or hemiparesis condition > 3 months;
* stroke-induced clinical deficits affecting motor, perceptual, or language functions, with NIHSS of 5-15;
* stroke in the middle cerebral artery territory;
* subjects able to understand, sign and date the informed consent form

Exclusion Criteria:

* non-ischemic mechanism, subarachnoid hemorrhage, primary intracerebral or intraventricular hemorrhage;
* pregnant or lactating women;
* alcohol or drug abuse in previous 3 months;
* significant medical diseases or infections;
* current participation in another investigational study or taking any investigational drug within last 4 weeks before the screening;
* unavailability of HLA-matched umbilical cord blood unit;
* investigator suggests that the subject would not suitable to perform the surgery or participate in the study

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-10; Primary Completion 2018-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale | 18 months, up to 36 months
  The change from the baseline in National Institutes of Health Stroke Scales

SECONDARY OUTCOMES:
European Stroke Scale (ESS) | 18 months, up to 36 months if applicable
  The change from baseline in ESS
Barthel Index | 18 months
Min-Mental State Examination (MMSE) | 18 months
  The change from baseline in MMSE
MRI | 18 months
  The change in MRI between pre-treatment and post-treatment

OTHER OUTCOMES:
Safety as assessed by the incidence and severity of adverse events, clinically-significant changes in lab tests, vital signs, physical and neurological examinations. | 18 months, up to 36 months follow-up
  Safety are assessed by the incidence and severity of adverse events, clinically-significant changes in lab tests, vital signs, physical and neurological examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Waisang Poon, MD, Principal Investigator — The Chinese University of Hong Kong, Prince of Wales Hospital; Gilberto Ka Kit Leung, MD, Principal Investigator — The University of Hong Kong, Queen Mary Hospital
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin